CLINICAL TRIAL: NCT06820710
Title: Multidomain Interventions to Improve the COgnitive and fUNctional Well-being of Elderly Individuals in Residential sTructures (I-COUNT)
Brief Title: Multidomain Interventions for Elderly Individuals in Residential Structures
Acronym: I-COUNT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Neuroscienze Consiglio Nazionale delle Ricerche (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2024-SPERIM_ALTRO-CR4; 5982/U6/24 (Other: CET Area Centro-Est Veneto)
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Aging; Age-Related Cognitive Decline; Sarcopenia; Long Term Care Facility; Cognitive Training; Physical Exercise; Functional Food; Nutritional Intervention; Vaccinations
Keywords: aging; long term care facilities; multidimensional interventions; cognitive training; physical exercise; nutritional intervention; functional foods; vaccinations
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise; Vaccination

STUDY DESIGN:
Intervention Model Description: Participants in the "experimental group: multidomain intervention" will undergo the planned interventions for a 6-month period, including physical activity and cognitive training; they will be offered to receive appropriate vaccinations according to the national vaccination calendar, and will be offered functional foods.
  Participants in the "control group" will be asked to continue with their usual activities.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidomain Intervention group (Experimental): The 6-month intervention will include supervised physical exercises (each session will last 40 minutes, three times a week, with accelerometers and smartwatches to monitor the physical activity performed), and cognitive stimulation (delivered by neuropsychologists twice a week for 30 minutes, in small groups). Participants in the intervention group will be advised to follow a Mediterranean diet, will receive functional foods (sourdough bread fortified with vegetable matrix rich in polyphenols and probiotic artichokes), and will be offered to receive appropriate vaccinations according to the national vaccination calendar.
  Interventions: Other: Physical activity; Other: Cognitive stimulation; Other: Nutritional Intervention; Other: Vaccinations
- Control group (usual activities) (No Intervention): Subjects in the control group will receive general information on healthy lifestyles and health, including risk factors.

INTERVENTIONS:
Other: Physical activity — Appropriate exercises for supervised small group sessions will be prescribed by a physiotherapist or expert in exercise science. Each session will last approximately 40 minutes, three times a week, and will be based on the international guidelines for physical exercise in the elderly population, and the VIVIFRAIL Multicomponent Physical Exercise Program to Prevent Frailty and the Risk of Falls. Accelerometers and other wearable sensors (smartwatches) will be used to monitor the physical activity performed.
  Arms: Multidomain Intervention group
Other: Cognitive stimulation — Cognitive stimulation will be delivered by expert neuropsychologists twice a week (48 sessions in total) for approximately 30 minutes. Residents will be divided into small groups (3-5 people) of similar cognitive level, and the intervention will be delivered using a computerized tool (REmote stimulation for COgnitive DEcline (RECODE) developed by researchers at the University of Padova with the aim of stimulating different domains (i.e., attention, working memory, visual memory, language, orientation and executive functions) through exercises of increasing difficulty.
  Arms: Multidomain Intervention group
Other: Nutritional Intervention — Participants in the intervention group will be advised to follow a Mediterranean diet and will also receive functional foods; in particular, they will be offered 80 g/day of sourdough bread fortified with vegetable matrix rich in polyphenols (e.g., olive leaves) and 100 g/day of probiotic artichokes on alternate days.
  Arms: Multidomain Intervention group
Other: Vaccinations — Participants in the intervention group will be offered to receive appropriate vaccinations according to the national vaccination calendar. Vaccine doses will be provided by the Department of Preventive Medicine, Vaccine Office, National Health Service, on prescription from the general practitioners.
  Arms: Multidomain Intervention group

SUMMARY:
The "Multidomain Interventions to improve the COgnitive and fUNctional well-being of elderly individuals in residential sTructures" (I-COUNT) study aims to test the feasibility and the effectiveness of a multidisciplinary intervention among elderly individuals living in long term care facilities (LTCFs). The intervention will include selected physical and cognitive training activities administered and monitored by new technologies, a dietary intervention including also functional foods, and the administration of vaccines according to the National plan. The multidomain intervention will last 6 months and will be compared with the standard care adopted in the same LTCFs.

DETAILED DESCRIPTION:
I-COUNT is a randomized controlled trial that will be conducted among residents in two residential facilities in Italy. Sixty participants will be enrolled in each residential facility (30 control group, 30 intervention group).

During the first phase of the study, eligible residents of the participating LTCFs will be enrolled according to the following inclusion and exclusion criteria. Baseline evaluations will be based on a geriatric multidimensional assessment including body composition assessment, physical performance assessment, Mediterranean diet adherence assessment, psychological and neuropsychological evaluations. Blood, plasma, stool and urine samples will also be collected.

In phase two, which will last 6 months, participants in the intervention group will undergo the planned interventions, while controls will be asked to continue with their usual activities. The physical activity will consist of three 40-minutes sessions per week, with personalized exercises prescribed by a physiotherapist and performed in small groups, under supervision. The cognitive training will be based on the computer program Remote stimulation for Cognitive Decline (RECODE), developed by the Department of General Psychology, University of the Padua, with two sessions per week. The intervention group will also receive functional foods (sourdough bread enriched with a vegetable matrix rich in polyphenols (olive leaves) and vegetables enriched with probiotics (artichokes)).

In phase 3, participants will be reassessed at 3 months (gut microbiota only), and 6 and 9 months after the start of the intervention (selected biomarkers, nutritional and anthropometric status, psychological health, physical performance tests, cognitive function, acceptability of the technological monitoring and interventions).

ELIGIBILITY:
Inclusion Criteria:

* age ≥70 years;
* resident in the identified LTCFs for at least 6 months;
* able to communicate and collaborate with the research team;
* Mini-Mental State Examination-MMSE ≥18.

Exclusion Criteria:

* estimated length of stay in the LTCFs<6 months;
* estimated life expectancy <6 months;
* previous gastrectomy or colectomy;
* presence of a nasogastric tube or percutaneous endoscopic gastrostomy (PEG);
* presence of dysphagia;
* inability to undergo psychometric tests for any reason;
* history of psychiatric illness according to clinical anamnesis;
* inability to walk.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the multidomain intervention on the gut microbiota composition | Baseline and 3 months after the start of the intervention
  Changes in gut microbiota biodiversity measured as species richness (number of different taxa identified in each sample) in the intervention group compared to control group
Effect of the multidomain intervention on the gut microbiota composition | Baseline and 3 months after the start of the intervention
  Changes in gut microbiota in term of the most represented bacterial taxa (such as Faecalibacterium prausnitzii, Akkermansia muciniphila, Bifidobacterium spp, Lactobacillus spp; measured as average relative abundance) in the intervention group compared to control group
Effect of the multidomain intervention on the gut microbiota composition | Baseline and 3 months after the start of the intervention
  Changes in gut microbiota in terms of gene or transcript counts (measured as counts) in the intervention group compared to control group

SECONDARY OUTCOMES:
Feasibility of the multidomain intervention | At the end of the intervention (6 months after the start)
  Number of drop out (number) in the intervention group compared to control group
Effect of the multidomain intervention on the gut microbiota composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in gut microbiota biodiversity measured as species richness (number of different taxa identified in each sample) in the intervention group compared to control group
Effect of the multidomain intervention on the gut microbiota composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in gut microbiota in terms of gene or transcript counts (measured as counts) in the intervention group compared to control group
Effect of the multidomain intervention on the gut microbiota composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in gut microbiota in term of the most represented bacterial taxa (such as Faecalibacterium prausnitzii, Akkermansia muciniphila, Bifidobacterium spp, Lactobacillus spp; measured as average relative abundance) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in cholesterol (measured in mg/dl) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in triglycerides (measured in mg/dL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in blood glucose (measured in mg/dL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in vitamin D (measured in nmol/L) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in transferrin (measured in mg/dL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in albumin (measured in g/dL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in FT3 (measured in pg/mL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers | Baseline, 6 and 9 months after the start of the intervention
  Changes in FT4 (measured in ng/dL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in IL-6 (measured in pg/mL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in BDNF (measured in ng/ml) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in s-RAGE (measured in pg/mL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in irisin (measured in ng/ml) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in IGF1 (measured in ng/mL) in the intervention group compared to control group
Effect of the multidomain intervention on specific biomarkers of aging | Baseline, 6 and 9 months after the start of the intervention
  Changes in ghrelin (measured in pg/mL) in the intervention group compared to control group
Effect of the multidomain intervention on the nutritional status | Baseline, 6 and 9 months after the start of the intervention
  Changes in Mini Nutritional Assessment (MNA, score 0-30, a higher score indicates a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on anthropometric status and body composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in body mass index (BMI, with weight measured in kg and height measured in m combined to report BMI in kg/m^2) in the intervention group compared to control group
Effect of the multidomain intervention on anthropometric status and body composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in waist circumference (measured in cm) in the intervention group compared to control group
Effect of the multidomain intervention on anthropometric status and body composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in calf circumference (measured in cm) in the intervention group compared to control group
Effect of the multidomain intervention on anthropometric status and body composition | Baseline, 6 and 9 months after the start of the intervention
  Changes in mid-upper arm circumference (measured in cm) in the intervention group compared to control group
Effect of the multidomain intervention on upper limb strength | Baseline, 6 and 9 months after the start of the intervention
  Changes in upper limb strength evaluated with electronic hand dynamometers (measured in kg) in the intervention group compared to control group
Effect of the multidomain intervention on general and domain-specific cognitive functioning | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Addenbrooke's Cognitive Examination (ACE-R, minimum 0, maximum 10, a higher score indicate a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on physical performance | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Short Physical Performance Battery (SPPB, minimum 0, maximum 12, a higher score indicates a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on psychological health | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Geriatric Depression Scale (GDS, minimum score 0, maximum score 30, a higher score indicates a worse outcome) in the intervention group compared to control group
Effect of the multidomain intervention on psychological health | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Perceived Stress Scale (PSS, minimum score 0, maximum score 40, a higher score indicates worse outcome) in the intervention group compared to control group
Effect of the multidomain intervention on psychological health | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Depression Anxiety Stress Scale (DASS-21, minimum score 0, maximum score 63, a higher score indicates worse outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Physical Health, minimum score 0, maximum score 100, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Psychological Health, minimum score 0, maximum score 100, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Social Relationships, minimum score 0, maximum score 100, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Environment, minimum score 0, maximum score 100, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Quality of Life, minimum score 0, maximum score 5, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on quality of life | Baseline, 6 and 9 months after the start of the intervention
  Changes in the World Health Organization Quality of Life Scale (WHOQOL-BREF Health Satisfaction, minimum score 0, maximum score 5, a higher score represents a better outcome) in the intervention group compared to control group
Effect of the multidomain intervention on sleep quality | Baseline, 6 and 9 months after the start of the intervention
  Changes in the Pittsburgh Sleep Quality Index (PSQI, minimum score 0, maximum score 21, a higher score indicates a worse outcome) in the intervention group compared to control group
Effect of the multidomain intervention on the number of hospitalization | 6 and 9 months after the start of the intervention
  Incidence (number) of hospitalizations during follow-up in the intervention group compared to control group
Effect of the multidomain intervention on the number of falls | 6 and 9 months after the start of the intervention
  Incidence (number) of falls during follow-up in the intervention group compared to control group

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - RSA Cremona Solidale, Cremona, Italy
  - AltaVita IRA, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romeo Z, Macchia E, Ceolin C, Devita M, Morandi A, Noale M, Maggi S; I-COUNT Study Group. Feasibility and Potential Effects of Multidomain Interventions to Improve the Cognitive and Functional Well-Being of Elderly Individuals in Residential Structures: The I-COUNT Pilot Study Protocol. Healthcare (Basel). 2025 Aug 14;13(16):1999. doi: 10.3390/healthcare13161999. PMID 40868616